CLINICAL TRIAL: NCT05016739
Title: Use of CADISS Medical Device to Facilitate Dissection of Epidural Fibrosis in Patients Who Undergo Revision in Spine Surgery After at Least One Year (CADISS1701)
Brief Title: Use of CADISS Medical Device to Facilitate Dissection of Epidural Fibrosis in Revision Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AuXin Surgery SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CADISS 1701
Record Dates: First submitted 2021-08-09; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Spine Surgery
Keywords: spine; lumbar; surgery; revision; CADISS; fibrosis; chemically assisted dissection
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CADISS System (Experimental)
  Interventions: Device: CADISS

INTERVENTIONS:
Device: CADISS — The CADISS® device was procured from AuXin Surgery. It consists in three elements:
  1. A single use disposable Remote Kit, containing a sterile cartridge, which prepares the Drug Product immediately before use, and the sterile tubing for fluid connexion. The Drug Product is a 30 ml sterile 5% mesna solution of pH 7.3+/-0.5
  2. Reusable stainless steel non-cutting mechanical instruments similar to those used in the normal practice, except for the provision of an internal irrigation channel bringing the Drug Product at the working edge.
  3. A pedal controlled electric motor driving the peristaltic cassette included in the disposable tubing in order to control the dispensing of the Drug Product during the procedure.

SUMMARY:
The CADISS® System, Chemically Assisted mechanical DISSection, is intended for the selective detachment of pathological tissue layers and/or fibrotic tissues in various surgical procedures without using cutting instruments. It is based on the property of the drug mesna (Sodium 2-mercaptoethane sulfonate) to cleave the disulfide bonds responsible for the adherence of pathological tissues and for the strength of fibrosis. Revision spine surgery is more difficult than primary surgery because of the development of fibrosis and scar tissues since the first operation. Fibrosis may develop in the spinal canal and will adhere strongly to the dura mater and to the nerve roots. This study is a prospective, multi-sites, open label, single cohort clinical trial evaluating the use of CADISS medical devices to facilitate dissection of epidural fibrosis in patients who undergo a revision in spine surgery after at least one year.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, weight > 30 Kg
* Eligible for Spine revision surgery, at least one year after primary surgery
* Agree to participate and sign the informed consent

The age and weight of patient are defined according to the instruction for use of the CADISS System currently on the EU market.

Exclusion Criteria:

* < 18 years old
* Weight ≤ 30 kg
* Primary surgery
* Known hypersensibility to mesna
* Patient is pregnant, breastfeeding or has wish of pregnancy during the study.
* Unable to sign the informed consent
* Participation in any study involving an investigational drug or device within the past 3 Months.
* Individuals under tutorship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Ability of the CADISS® System to dissect fibrosis without cutting | Surgery
  Percentage of successful dissection

SECONDARY OUTCOMES:
Global satisfaction score when using the | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice
The facilitation of fibrosis detachment with the CADISS System | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice
The reduction of bleeding with the use of the CADISS System | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice
The capability of the CADISS system to highlights cleavage plane | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice
The speed of action of the mesna solution after local instillation | Surgery
  Likert scale - 0 to 10. A score of 0 representing the worse outcome
The ease of use of the CADISS System | Surgery
  Likert scale - 0 to 10. A score of 0 representing the worse outcome
The easy of control of the topical application with the CADISS System | Surgery
  Likert scale - 0 to 10. A score of 0 representing the worse outcome
Adverse events | surgery, at hospital discharge minimum 1 day after surgery, 6 weeks
  All CADISS related Adverse events will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse Lubansu, MD, Principal Investigator — University Hospital Erasme, Brussels, Belgium
Locations (1):
- AuXin Surgery, Louvain-la-Neuve, Belgium